CLINICAL TRIAL: NCT02744820
Title: A Double Blind, Placebo-controlled, Randomised, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GMC-252 in Healthy Male Subjects and Male Type 2 Diabetics
Brief Title: Multiple Ascending Dose Study of GMC-252-L-Lys Salt in Healthy Subjects and Type 2 Diabetics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It was considered by the sponsor that the study objective has been met by dosing 13 instead of 15 patients
Sponsor: Genmedica Therapeutics S.L. (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMC-252-1.03
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Part 1) (Placebo Comparator): Multiple ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Salt Other: Placebo
  Interventions: Drug: GMC-252-L-Lysine Salt; Other: Placebo
- Cohort 2 (Part 1) (Placebo Comparator): Multiple ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Salt Other: Placebo
  Interventions: Drug: GMC-252-L-Lysine Salt; Other: Placebo
- Cohort 3 (Part 1) (Placebo Comparator): Multiple ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Salt Other: Placebo
  Interventions: Drug: GMC-252-L-Lysine Salt; Other: Placebo
- Cohort 4 (Part 2) (Placebo Comparator): Multiple ascending oral administrations of GMC-252-L-Lysine Salt and matching placebo
  Interventions:
  Drug: GMC-252-L-Lysine Salt Other: Placebo
  Interventions: Drug: GMC-252-L-Lysine Salt; Other: Placebo

INTERVENTIONS:
Drug: GMC-252-L-Lysine Salt — 1 dose by oral route, once a day, 28 days
  Other Names: GMC-252-L-Lys Salt
Other: Placebo — Matching doses by oral route, once a day, 28 days

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of multiple oral doses of GMC-252-L-Lysine salt (GMC-252) in healthy subjects and type 2 diabetics.

The secondary objective is to explore the effect of multiple oral doses of GMC-252 on pharmacodynamic(PD) parameters in type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria

Part 1 (Healthy Subjects) and Part 2 (Type 2 Diabetic Patients):

1. Diet: Able to eat standard food, no vegetarians.
2. Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.
3. Consent: Demonstrates understanding of the study and has given signed, voluntary written informed consent.
4. Have no known hypersensitivity to diflunisal, NAC or other NSAIDs.
5. No history of blood diseases including but not limited to clinically significant platelet diseases and coagulation abnormalities.
6. No clinically relevant gastrointestinal disease.
7. Have an estimated creatinine (CREA) clearance>70 mL/min/surface area (CREA clearance will be calculated from the serum CREA value by using the Cockroft and Gault formula).
8. Have no history of heart failure or uncontrolled hypertension or other known clinically significant cardiovascular disease.
9. Have no history of bronchial asthma or 'Aspirin Triad' (chronic rhino-sinusitis with polyps, severe asthma and intolerance to aspirin or other NSAIDs).
10. Have no clinically significant abnormality of liver tests before entry into the study.
11. A negative urinary drugs of abuse screen, determined within 28 days before the first dose (N.B. a positive alcohol result may be repeated at the discretion of the Investigator).
12. Negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
13. No clinically significant abnormalities in a 12-lead ECG determined within 28 days before the first dose.
14. No history of clinically significant renal disease or any food intolerance.
15. Willing to use 2 effective methods of contraception i.e. established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months afterwards.

Additional Criteria for Part 1 (Healthy Subjects):

1. Healthy males aged 18 to 55 inclusive.
2. Body mass index (BMI) within the range of 18-30 kg/m2 inclusive.
3. Non-Smokers (including e-cigarettes) who have abstained from smoking for at least 6 months.

Additional Criteria for Part 2 (Type 2 Diabetic Patients):

1. Males aged 18 to 65 inclusive. BMI within the range of 18-38 kg/m2 inclusive.
2. Diagnosis of T2DM according to the World Health Organization criteria.
3. HbA1c between 7.0% and 12.0 % inclusive.
4. Currently treated with metformin with a stable treatment regimen for 3 months or more prior to the Screening Visit, and not receiving other anti-diabetic medications. Allowed medication during the study include metformin, statin (3-hydroxy-3-methylglutaryl-coenzyme A (HMG CoA) reductase inhibitors), paracetamol up to 3 g/day, low doses of aspirin and antihypertensive drugs if the doses are not changed in the 3 months before the start of screening. Other allowed medications will be approved by PI and Sponsor before a patient can be enrolled. Diflunisal (a test drug component) may decrease the antihypertensive activityof many of the currently used antihypertensive medications, such as β-blockers, alpha (α)-blockers, loop diuretics, angiotensin converting enzyme (ACE inhibitors), angiotensin 2 receptor blockers, calcium channel blockers. Therefore, patients who are on current stable antihypertensive medications will be subjected to close monitoring of their blood pressure throughout the study.
5. Stable dietary habits and regimen of treatment for concomitant diseases for 1 month or more prior to the Screening Visit.
6. Subject able and willing to undergo oral glucose tolerance test (OGTT).

Exclusion Criteria

Part 1 (Healthy Subjects) and Part 2 (Type 2 Diabetic Patients):

1. A clinically significant history of previous allergy / sensitivity to any of the GMC-252 components, NAC or diflunisal.
2. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
3. Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
4. Donation of 450 mL or more blood within the previous 3 months.
5. A clinically significant history of drug, alcohol or other substance abuse in the past 2 years.

Additional Criteria for Part 1 (Healthy Subjects):

1. A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Receipt of regular medication within 28days of the first dose that may have an impact on the safety and objectives of the study (at the Investigator's discretion).
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.

Additional Criteria for Part 2 (Type 2 Diabetic Patients):

1. Diagnosis/General Health:

   * Diabetic autonomic or sensory neuropathy including gastroparesis, diabetic nephropathy or untreated active proliferative retinopathy.
   * Clinically significant abnormalities in laboratory evaluation (including clinical biochemistry, haematology and urinalysis) in the opinion of the Investigator.
2. Diseases:

   * Uncontrolled hypertension (blood pressure ≥ 160/100 mmHg), severe or unstable angina, coronary insufficiency, congestive heart failure, clinically significant (in the opinion of the Investigator) renal or hepatic disease.
   * Previous gastric or intestinal surgerythat might impact drug absorption.
   * Malignancy within 5 years of the start of the study, except for successfully treated local basal cell carcinoma
   * Current or relevant previous history, of clinically significant psychiatric illness.
3. Medications:

   * Current use of insulin or any previous use of insulin other than as part of a clinical trial or associated with surgical procedure or acute illness for up to 7 days.
   * Use of any anti diabetic medication other than metformin in the 3 months prior to study entry.
   * Current use of any anticoagulant drug e.g. warfarin, heparin.
   * Prior use (within 48 h of dosing) of any drug that could have altered gastric motility (domperidone, cyclizine, metoclopramide, prochlorperazine), or cholestyramine.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 28 days plus 14 days post last dose
  Physical status (Vital signs; 12-lead ECG; Urinalysis; Haematology and biochemistry)

SECONDARY OUTCOMES:
Maximal Concentration (Cmax) | 28 days plus 14 days post last dose
Area Under the Concentration-Time Curve | 28 days plus 14 days post last dose
Time to reach steady state | 28 days plus 14 days post last dose

OTHER OUTCOMES:
Preliminary effect on Fasting blood glucose (Cohort 4 only) | 28 days plus 14 days post last dose
Preliminary effect on oral glucose tolerance test (OGTT) (Cohort 4 only) | 28 days plus 14 days post last dose
Preliminary effect on Insulin levels (Cohort 4 only) | 28 days plus 14 days post last dose
  Insulin
Preliminary effect on C-Peptide levels (Cohort 4 only) | 28 days plus 14 days post last dose
Preliminary effect on Fructosamine levels (Cohort 4 only) | 28 days plus 14 days post last dose
Preliminary effect on %HbA1c (Cohort 4 only) | 28 days plus 14 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams, MBBS, Principal Investigator — Simbec Research
Locations (2):
- United Kingdom (2):
  - BioKinetic Europe Ltd., Belfast
  - Simbec Research Ltd, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: Undecided